CLINICAL TRIAL: NCT04771663
Title: Variability of SpO2 Measurements Depending on the Choice of Finger for Sensor Placement
Acronym: FinSpO2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Czech Technical University in Prague (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CzechTU
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Hypoxia; Hypercapnia
MeSH Terms: conditions — Hypoxia; Hypercapnia

STUDY DESIGN:
Intervention Model Description: Interventional single blinded randomized crossover prospective study
Who Masked: Participant
Masking Description: The participant undergoes two phases of the experiment and the participant does not know which one
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypoxic (Experimental): In this phase, participants inhale the hypoxic mixture for five minutes.
  Interventions: Other: Breathing a mixture of O2, N2 and CO2 and monitoring SpO2 on each finger
- Hypoxic and Hypercapnic (Experimental): In this phase, participants inhale the hypoxic and hypercapnic mixture for five minutes.
  Interventions: Other: Breathing a mixture of O2, N2 and CO2 and monitoring SpO2 on each finger

INTERVENTIONS:
Other: Breathing a mixture of O2, N2 and CO2 and monitoring SpO2 on each finger — The experiment consists of two separate phases. In one phase, the volunteers inhale one of the mixtures for five minutes. After enough time of recovery, the volunteers undergo the other phase in which they inhale the other mixture of gases. Both phases of the measurement will begin with a two-minute stabilization phase, during which the physiological values of the volunteer will be checked. During the experiment, non-invasive SpO2 measurements will be performed continuously on the individual fingers of both volunteer hands throughout the experiment.

SUMMARY:
The aim of the project is to experimentally determine the effect of the choice of finger for the placement of a pulse oximeter sensor on the results of measuring peripheral blood oxygen saturation (SpO2) in a healthy person with short-term hypoxia and hypercapnia.

DETAILED DESCRIPTION:
The aim of the project is to experimentally determine the effect of the choice of finger for the placement of a pulse oximeter sensor on the results of measuring peripheral blood oxygen saturation (SpO2) in a healthy person with short-term hypoxia and hypercapnia. This is an intervention prospective study that will take place at the Faculty of Biomedical Engineering, especially on FBMI students. The experiment consists of two phases, in which in the first phase, the volunteers will inhale the hypoxic mixture for five minutes after the stabilization phase. In the second phase, volunteers inhale a hypoxic and hypercapnic mixture. During the experiment, non-invasive SpO2 measurements will be performed continuously on individual fingers of both volunteer hands.

ELIGIBILITY:
Inclusion Criteria:

* Passing the initial examination, which will determine the following data: finger circumference, heart rate, blood pressure and blood oxygen saturation

Exclusion Criteria:

* post-traumatic conditions of the upper limbs affecting the perfusion of the fingers or injuries or skin diseases on the fingers.
* pneumothorax or a condition after cardiovascular surgery.
* anemia, bradycardia, hemoglobinopathy or other diseases of the cardiovascular system, pregnancy, diabetes, hypotension or hypertension.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-10 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
Does it depend on which finger is the sensor placed for SpO2 values? | Up to 12 weeks
  The experiment can help determine if it depends on which finger the finger sensor will be placed to measure SpO2. Appropriate finger selection for SpO2 measurements could help to better interpret the measured values and possibly increase the success in diagnosing health events.

CONTACTS AND LOCATIONS:
Overall Officials: Karel Roubík, Study Director — Czech Technical University in Prague, FBMI
Locations (1):
- Czech Technical University in Prague, Kladno, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rafl J, Kulhanek F, Kudrna P, Ort V, Roubik K. Response time of indirectly accessed gas exchange depends on measurement method. Biomed Tech (Berl). 2018 Nov 27;63(6):647-655. doi: 10.1515/bmt-2017-0070. PMID 28802098